CLINICAL TRIAL: NCT06050226
Title: A Multi-center, Randomized, Open-label, Phase 2 Study to Evaluate the Efficacy and Safety of MY008211A Tablets in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria and Active Hemolysis.
Brief Title: A Study of MY008211A in Adult Patients With Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wuhan Createrna Science and Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MY008211A-PNH-2-01
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2023-09

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm1：low MY008211A dose (Experimental): Participants will receive low MY008211A dose orally b.i.d
  Interventions: Drug: MY008211A tablets
- Arm2：high MY008211A dose (Experimental): Participants will receive high MY008211A dose orally b.i.d
  Interventions: Drug: MY008211A tablets

INTERVENTIONS:
Drug: MY008211A tablets — The first 10 participants will be received low-dose MY008211A tablets, and the next 30 participants will be randomized to low-dose or high-dose treatment arms in a 1:2 ratio.
  Other Names: MY008211A

SUMMARY:
The main purpose of this study is to evaluate the efficacy of MY008211A in adult patients with PNH , showing signs of active hemolysis, in China.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether MY008211A is efficacious and safe for the treatment of PNH patients who are naive to complement inhibitor therapy, including anti-C5 antibody.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ≥ 18 years of age, BMI≥18 kg/m2，with a diagnosis of PNH confirmed by laboratory tests, according to the PNH diagnostic criteria in the Chinese Guidelines for the Diagnosis and Treatment of Rare Diseases (2019 edition) , and flow cytometry with clone size ≥ 10%.
* Mean hemoglobin level <100 g/L.
* LDH > 1.5 x Upper Limit of Normal (ULN)
* Vaccination against Neisseria meningitidis infection is required prior to the start of study treatment. If not received previously, vaccination against Streptococcus pneumoniae and Haemophilus influenzae infections should be given.

Exclusion Criteria:

* Patients with reticulocytes <100x10^9/L; platelets <30x10^9/L; neutrophils <0.5x10^9/L.
* Were using a complement inhibitor before the first administration of MY008211A tablets or had discontinued a previous complement inhibitor for less than five half-lives or 120 days, whichever was the longest.
* History of recurrent invasive infections caused by encapsulated organisms, e.g. meningococcus or pneumococcus.
* Known or suspected hereditary complement deficiency
* Previous bone marrow or hematopoietic stem cell transplantation.
* Previous splenectomy.
* A history of malignancy within 5 years before screening, except cured local basal cell carcinoma of the skin and carcinoma in situ of the cervix.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving a sustained increase in hemoglobin levels of ≥ 20 g/L in the absence of red blood cell transfusion. | up to 84 days
  Proportion of participants achieving a sustained increase from baseline in hemoglobin levels of ≥ 20 g/L assessed , in the absence of red blood cell transfusions

SECONDARY OUTCOMES:
Proportion of participants achieving sustained hemoglobin levels ≥ 120 g/L in the absence of red blood cell transfusions. | up to 84 days
  Proportion of participants achieving sustained hemoglobin levels ≥ 120 g/L in absence of red blood cell transfusion
Change from baseline in hemoglobin concentration. | up to 84 days
  Change from baseline in hemoglobin concentration (g/L) in absence of red blood cell transfusion
Change from baseline in serum LDH levels. | up to 84 days
  Change from baseline in serum LDH levels (U/L)
Change from baseline in Reticulocyte count. | up to 84 days
  Change from baseline in Reticulocyte count (×10^9/L)
Changes from baseline in transfusion volume. | up to 84 days
  The average number of red blood cells transfused per week
Change in the level of PNH red cell clones. | up to 84 days
  Change from baseline in the level of PNH red cell clones.
Occurrences of AEs occurring between Day 1 and Day 84. | up to 84 days
  Adverse Events (AEs)

OTHER OUTCOMES:
Changes from baseline in alternative complement pathway activity. | up to 84 days
  Alternative complement pathway activity measured by the WIESLAB® kit.
Change from baseline in plasma levels of the Bb fragment. | up to 84 days
  Bb fragment cleaved by factor B of complement.
Maximum Plasma Concentration (Cmax) Of MY008211A tablets | up to 84 days
  PK parameters
Area Under The Concentration Versus Time Curve (AUC) Of MY008211A | up to 84 days
  PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: Fengkui Zhang, Ph.D, Principal Investigator — Blood Disease Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Disease Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality, China